CLINICAL TRIAL: NCT03372018
Title: Promotora Intervention for Metabolic and Mental Health
Brief Title: Promotora-Led Intervention for Metabolic and Mental Health
Acronym: PRIME2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Matthew J O'Brien, Assistant Professor of Medicine and Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00202244; R03DK109243 (NIH)
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: PreDiabetes; Obesity; Metabolic Disease; Body Weight Changes; Diabetes Mellitus
MeSH Terms: conditions — Prediabetic State; Obesity; Metabolic Diseases; Body Weight Changes; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promotora-led intervention (PLI) (Experimental): PLI -DPP protocol was developed from original DPP materials and culturally tailored for the target population based on formative research. The core PL-DPP curriculum includes 14 group sessions of 90 minutes duration. One promotora will lead each session in Spanish using behavioral strategies to discuss lifestyle behaviors, exploring such topics as being active, low-fat diets, portion control, self monitoring, problem solving and life-style changes.
  Interventions: Behavioral: Promotora-led Intervention (PLI)
- Usual care (UC) (Active Comparator): UC participants will receive standard educational materials in Spanish discussing mental health and diabetes prevention. UC participants will be encouraged to continue all routine medical care during the study.
  Interventions: Behavioral: Usual care (UC)

INTERVENTIONS:
Behavioral: Promotora-led Intervention (PLI) — Behavioral life-style program with cognitive-behavioral content lead by a team of trained community health workers (called promotoras) with the following principal goals - encouraging participants to lose 7% of their total weight and complete 150 minutes of moderate physical activity per week.
  Arms: Promotora-led intervention (PLI)
Behavioral: Usual care (UC) — Participants in this arm will be given educational materials in spanish discussing mental health and diabetes prevention.
  Arms: Usual care (UC)

SUMMARY:
Evidence-based programs to prevent diabetes among high-risk individuals are less effective among those who also have mental health needs. This study involves developing and pilot testing the first adaptation of the landmark Diabetes Prevention Program lifestyle intervention to simultaneously treat prediabetes and elevated mental health symptoms. This project has large potential to impact public health, given that more than half of the U.S. adult population has either of these conditions, and is at risk for developing comorbid diabetes and mental illness.

DETAILED DESCRIPTION:
The overall goal of this study is to develop an effective and potentially scalable intervention to prevent diabetes in people with elevated mental health symptoms (EMS) and prediabetes. This study focuses on Latinos, a demographic group at particularly high risk for these related conditions. Experience from the Diabetes Prevention Program (DPP), and related translational studies, suggests that the evidence-based DPP lifestyle intervention is less effective among depressed individuals. The proposed Promotora Intervention for Metabolic and Mental Health (PRIME2) will be the first adaptation of the DPP lifestyle intervention to simultaneously address mental health and prediabetes in a program delivered by promotoras, or community health workers.

ELIGIBILITY:
Inclusion Criteria:

* Latino ethnicity
* Spanish fluency
* Age ≥18 years
* BMI ≥25 kg/m2
* And "increased risk of diabetes" (ADA Diabetes Risk Score ≥5 as determined by 7-item questionnaire and/or hemoglobin A1C ≥ 5.7%)

Exclusion Criteria:

* Hemoglobin A1C ≥ 6.5%
* Current or planned pregnancy during the study period
* Chronic conditions that could affect potential participants' ability to participate (osteoarthritis, heart disease, pulmonary disease requiring oxygen or daily bronchodilator use, and severe psychiatric disease)
* Medical comorbidities that could influence weight loss or weight gain (thyroid disease, cancer, and HIV)
* Medications that could affect weight or glucose metabolism (thiazide diuretics, β-blockers, and systemic glucocorticoids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 months
  Weight change from baseline.

SECONDARY OUTCOMES:
Perceived Stress | 3 months
  The Perceived Stress Scale (PSS) is a 14-item tool meant to measure how different situations affect participant feelings and perceived stress. Individual scores on the PSS range from 0 to 40 with higher scores indicating higher perceived stress. Each item is rated on a 5-point scale ranging from never (0) to almost always (4).The total score reported for each participant.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Cardiometabolic marker - A1C | 3 months
  Hemoglobin A1C change from baseline measured from a fingerstick capillary blood sample using a DCA 2000/Vantage portable analyzer.
Cardiometabolic marker - waist circumference | 3 months
  Waist circumference change from baseline assessed using a measuring tape around the top of the iliac crests at end-expiration.
Beck Depression Inventory | 3 months
  levated depressive symptoms were assessed using the Beck Depression Inventory (BDI), a depression screening instrument. The BDI score recorded at the enrollment visit will be considered the baseline BDI score. The last measured BDI score within 3 months after the baseline visit is the follow-up score used to calculate mean BDI change.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, MD, MSc, Principal Investigator — Assistant Professor of Medicine and Preventive Medicine
Locations (1):
- Northwestern Univeristy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No